CLINICAL TRIAL: NCT06937385
Title: Randomized, Prospective, Open-label, Controlled Trial of 0.5% Bupivacaine Lower Cervical Intramuscular Injection vs IV Medications in Treatment of Non-Traumatic Headache in the Emergency Department
Brief Title: 0.5% Bupivacaine Lower Cervical Intramuscular Injection vs IV Medications for Headache Treatment
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: HCA Florida North Florida Hospital (Other)
Responsible Party: Principal Investigator, Zhengqiu Zhou, Faculty, HCA Florida North Florida Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-302
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Headache; Migraine; Tension Headache; Occipital Neuralgia
Keywords: headache; bupivicaine; cervical injection; paraspinous injection
MeSH Terms: conditions — Headache; Migraine Disorders; Tension-Type Headache | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous medication (Active Comparator): physicians choice of intravenous medication for headache treatment
  Interventions: Drug: standard IV treatment for headache
- cervical IM injection (Experimental): bilateral cervical injections of 0.5% bupivacaine into the paraspinous muscle at the c6-7 location
  Interventions: Drug: 0.5% Bupivacaine HCl

INTERVENTIONS:
Drug: 0.5% Bupivacaine HCl — bilateral cervical injections of 0.5% bupivacaine into the paraspinous muscle at the c6-7 location for headache treatment
  Other Names: cervical IM injection
  Arms: cervical IM injection
Drug: standard IV treatment for headache — physicians choice of IV medications in treatment of headache
  Arms: Intravenous medication

SUMMARY:
Headache is a frequent chief complaint among patients presenting to the Emergency Department (ED), accounting for 2.1 million visits annually in the United States. Often, individuals resort to ED care only after over-the-counter or home remedies have failed, leading to the predominant use of intravenous (IV) medications in the ED, including NSAIDs, triptans, neuroleptics, antiepileptics, and dopaminergic antagonists. Unfortunately, these pharmacologic treatments frequently induce side effects such as cognitive impairment, extrapyramidal reactions, and the potential for medication dependency. In the ED, patients frequently require concurrent administration of multiple systemic medications to achieve satisfactory pain relief, thereby elevating the risk associated with medication use. Despite these medication regimens, a significant portion of patients continue to experience inadequate pain relief. Consequently, the search for an optimal headache therapy-characterized by rapid and effective pain relief, long lasting results, minimal side effects, and allows for rapid ED patient turnover-continues to be a popular area of research in emergency medicine. The investigators plan to evaluate the use of 0.5% bupivacaine cervical IM injection at the c6-7 location for the treatment of non traumatic headaches using a non-inferiority design, randomized, prospective, open-label, controlled trial comparing it to physicians choice of intravenous medications in treatment of headache in the Emergency Department at North Florida Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient has to be able to provide own consent
* English-speaking only
* Non traumatic headache with VAS pain score of 5 or above out of 10

Exclusion Criteria:

* traumatic headache
* Confused patients
* allergy to bupivacaine
* infection over injection site
* recent neck surgery
* hemodynamically unstable
* bleeding disorder
* anticoagulation use
* pregnant, lactating women
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale pain score 0-10 | 24 hours
  Pain score at 30 minutes and 24 hours after treatment. 0 being no pain and 10 being the worse pain possible.

SECONDARY OUTCOMES:
Emergency department length of stay | 24 hours
  Duration that patients stayed in the Emergency department for
Need for additional medications | 24 hours
  Whether an additional medication was given to patients after 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Hoelle, MD, Principal Investigator — HCA north florida hospital emergency department
Locations (1):
- HCA Florida north florida Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared to protect patient safety and their healthcare information.